CLINICAL TRIAL: NCT00615316
Title: Guaraná ("Paullinia Cupana") for Radiation Related Fatigue in Breast Cancer Patients: Results Of A Pilot Double Blind Randomized Study
Brief Title: Guaraná for Radiation Related Fatigue in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Auro Del Giglio, MD, Chairman of Oncology and Hematology, Faculdade de Medicina do ABC
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 365/2006
Record Dates: First submitted 2008-02-04; First posted 2008-02-14 (Estimated); Last update posted 2008-02-14 (Estimated); Status verified 2008-02

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Guaraná
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guaraná — Guaraná extract 75mg/day
  Other Names: Paullinia Cupana
  Arms: A
Drug: Placebo — Placebo 1tab/d
  Arms: B

SUMMARY:
We hypothesize that Guaraná, a native plant from the Amazon, might improve radiation-induced fatigue in breast cancer patients undergoing treatment. In order to assess this, we randomized patients to either guaraná extract or to placebo, switching the assigned treatment mid-term through the radiation.

DETAILED DESCRIPTION:
The aim of this study is evaluate the favourable effects of Guaraná in memory and cognition in humans After approval by our Institutional Review Board, we included consenting patients with a histological diagnosis of early stage Breast Cancer for whom adjuvant radiation therapy was indicated. We excluded patients with a previous history of Radiation Therapy, anemia or clinical depression. We also excluded patients who were unable to grant informed consent or those who had medical contraindindications for the use of Guaraná (because of its psycho stimulant effect) such as uncontrolled hypertension, previous history of cardiac arrhythmia and insomnia.

The radiation therapy for patients who underwent mastectomy consisted of 28 fractions of 180cGy.

This study had a double-blind randomized design with crossover between experimental arms. After getting informed consent, we randomized patients at the beginning of radiation treatments (Phase I) to either 75 mg of Guaraná extract daily (Group A) or to Placebo (Group B). Randomization was centralized by the pharmacist. Halfway through the radiation treatments (Phase II), we switched patients from placebo to guaraná and vice versa. The protocol ended at the last session of radiation treatments (Phase III). In each of these three phases a new assessment of fatigue and depressive symptoms was undertaken, ie: immediately before the first radiation treatment (phase I); at switching (phase II) and right before the start of the last radiation treatment (phase III). At these three assessment points, patients had to complete the Chalder Fatigue Scale,4 the MD Anderson Brief Fatigue Inventory (available at http://www.mdanderson.org/topics/fatigue/) available in Portuguese, and the Beck Inventory Depression Scale II also validated in Portuguese.

We conducted the statistical analysis of the data with the Numerical Control Software Solution (www.ncss.com). We employed the repeated measures analysis of variance (ANOVA) test to compare tests scores within the same patient group and the ANOVA test to compare test's scores between the two groups (at similar phases of the study).

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of early stage Breast Cancer
* 18 years old or older

Exclusion Criteria:

* prior breast radiation
* anemia
* clinical depression
* unable to sign informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Fatigue | 5 weeks

SECONDARY OUTCOMES:
Depression | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Auro Del Giglio, MD, PhD, Principal Investigator — ABC Foundation School of Medicine
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil